CLINICAL TRIAL: NCT04990531
Title: Low-fielD magnEtiC Resonance Imaging of pulmonarY Parenchyma Changes Associated wiTh Confirmed SARS-CoV-2 Infection in Children and Adolescents
Brief Title: Low-field Magnetic Resonance Imaging of Pediatric COVID-19
Acronym: DECRYPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 206_21 B
Record Dates: First submitted 2021-07-22; First posted 2021-08-04 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-07

CONDITIONS: Sars-CoV-2 Infection; Lung Fibrosis; Covid19
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 subjects (Experimental): Childrens and adolescent with PCR-proven previous SARS-CoV-2 infection
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Blood sample
- Healthy controls (Active Comparator): Healthy controls negative for previous SARS-CoV-2 infection
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Low-field magnetic resonance imaging — Imaging of lung parenchyma and function by LF-MRI
Diagnostic Test: Blood sample — Blood sample for diagnostic testing

SUMMARY:
SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) is a new coronavirus and identified causative agent of COVID-19 disease. They predominantly cause mild colds but can sometimes cause severe pneumonia. The long-term consequences are still largely unexplained and misunderstood, especially in children and adolescents. The aim of this study is to assess the frequency of pulmonary skeletal changes in pediatric and adolescent patients using low-field magnetic resonance imaging (LF-MRI) in the setting of proven past SARS-CoV-2 infection.

DETAILED DESCRIPTION:
SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) is a new coronavirus and identified causative agent of COVID-19 disease. They predominantly cause mild colds, but can sometimes cause severe pneumonia. While the molecular basis for the changes in lung tissue or multi-organ involvement has been described, the age-specific long-term consequences, especially in children and adolescents, are still largely unexplained and not understood. Early publications from the primarily affected Chinese provinces described rather mild, partly asymptomatic courses in children. This is consistent with the observation that the risk of severe COVID-19 disease increases steeply from the age of 70 years, and is also determined by the severity of obesity and other risk factors. Developmental expression of tissue factors may be one reason for the relative protection of younger patients from severe courses of the disease.

However, it is now becoming increasingly clear that some individuals with milder initial symptoms of COVID-19 may suffer from variable and persistent symptoms for many months after initial infection - this includes children. A modern low-field MRI is located in Erlangen, Germany. This technique has already been used to demonstrate persistent damage to lung tissue in adult patients after COVID-19. The device with a field strength of 0.55 Tesla (T) currently has the world's largest bore (and is thus particularly suitable for patients with claustrophobia, among other things), a very quiet operating noise, and lower energy absorption in the tissue due to the weaker magnetic field than MRI scanners with 1.5T or 3T. This allows MRI imaging in a very wide pediatric population without the need for sedation.

The purpose of this study is to assess the frequency of lung parenchymal changes using low-field magnetic resonance imaging (LF-MRI) in pediatric and adolescent patients with past SARS-CoV-2 infection detected by PCR.

ELIGIBILITY:
Covid-19 group

Inclusion Criteria:

* (Past) Positive SARS-CoV-2 Infection (PCR proven)
* Age 5 to <18 years

Exclusion Criteria:

* Acute SARS-CoV-2 Infection and Isolation
* Quarantine
* Pregnancy
* Critical Illness
* No consent to LF_MRI
* General contraindications for LF-MRI, such as electrical implants, pace makers, perfusion pumps)

Healthy controls

Inclusion Criteria:

- Age 5 to <18 years

Exclusion Criteria:

* (Past) Positive SARS-CoV-2 Infection (PCR or antigen test proven)
* Suspect for lung disease
* Acute respiratory infection/symptomatic
* Acute SARS-CoV-2 Infection and Isolation
* Quarantine
* Pregnancy
* Critical Illness
* No consent to LF_MRI
* General contraindications for LF-MRI, such as electrical implants, pace makers, perfusion pumps)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-12-29 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Low-field magnetic resonance imaging | Single time point (1 day)
  Lung parenchymal changes (Ground-glass opacification/opacity (GGO))

SECONDARY OUTCOMES:
Blood sample: Serum | Single time point (1 day)
  Antibodies against SarS-CoV-2 (spike proteine)
Blood sample: Serum | Single time point (1 day)
  Antibodies against SarS-CoV-2 (nuceleocapsid)
Blood sample: Leucocytes | Single time point (1 day)
  Physical properties of single cells: Deformation
Blood sample: Leucocytes | Single time point (1 day)
  Physical properties of single cells: Cells size [µm³]
Blood sample: Leucocytes | Single time point (1 day)
  Physical properties of single cells: Youngs modulus [kPa³]
Blood sample: Erythrocytes | Single time point (1 day)
  Physical properties of single cells: Deformation
Blood sample: Erythrocytes | Single time point (1 day)
  Physical properties of single cells: Cells size [µm³]
Blood sample: Erythrocytes | Single time point (1 day)
  Physical properties of single cells: Youngs modulus [kPa³]
Blood sample: Monocytes | Single time point (1 day)
  Physical properties of single cells: Deformation
Blood sample: Monocytes | Single time point (1 day)
  Physical properties of single cells: Cells size [µm³]
Blood sample: Monocytes | Single time point (1 day)
  Physical properties of single cells: Youngs modulus [kPa³]
Low-field magnetic resonance imaging | Single time point (1 day)
  Lung functional changes (Ventilation defects)
Low-field magnetic resonance imaging | Single time point (1 day)
  Lung functional changes (Perfusion defects)
Low-field magnetic resonance imaging | Single time point (1 day)
  Lung functional changes (Combined defects)
Blood sample: IL-6 | Single time point (1 day)
  Serum level of IL-6
Blood sample: C-reactive protein | Single time point (1 day)
  Serum level of C-reactive protein
Blood sample: D-dimers | Single time point (1 day)
  Serum level of D-dimers

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  Individual participant data will not be available Study Protocol and Statistical Analysis Plan will be available The data will be available beginning 9 months and ending 36 months following article publication.
  The data will be available to researchers who provide a methodologically sound proposal.
  The data will be available for individual participant data meta-analysis, only. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

REFERENCES:
- [Background] Sajuthi SP, DeFord P, Li Y, Jackson ND, Montgomery MT, Everman JL, Rios CL, Pruesse E, Nolin JD, Plender EG, Wechsler ME, Mak ACY, Eng C, Salazar S, Medina V, Wohlford EM, Huntsman S, Nickerson DA, Germer S, Zody MC, Abecasis G, Kang HM, Rice KM, Kumar R, Oh S, Rodriguez-Santana J, Burchard EG, Seibold MA. Type 2 and interferon inflammation regulate SARS-CoV-2 entry factor expression in the airway epithelium. Nat Commun. 2020 Oct 12;11(1):5139. doi: 10.1038/s41467-020-18781-2. PMID 33046696
- [Background] Ziegler CGK, Allon SJ, Nyquist SK, Mbano IM, Miao VN, Tzouanas CN, Cao Y, Yousif AS, Bals J, Hauser BM, Feldman J, Muus C, Wadsworth MH 2nd, Kazer SW, Hughes TK, Doran B, Gatter GJ, Vukovic M, Taliaferro F, Mead BE, Guo Z, Wang JP, Gras D, Plaisant M, Ansari M, Angelidis I, Adler H, Sucre JMS, Taylor CJ, Lin B, Waghray A, Mitsialis V, Dwyer DF, Buchheit KM, Boyce JA, Barrett NA, Laidlaw TM, Carroll SL, Colonna L, Tkachev V, Peterson CW, Yu A, Zheng HB, Gideon HP, Winchell CG, Lin PL, Bingle CD, Snapper SB, Kropski JA, Theis FJ, Schiller HB, Zaragosi LE, Barbry P, Leslie A, Kiem HP, Flynn JL, Fortune SM, Berger B, Finberg RW, Kean LS, Garber M, Schmidt AG, Lingwood D, Shalek AK, Ordovas-Montanes J; HCA Lung Biological Network. Electronic address: lung-network@humancellatlas.org; HCA Lung Biological Network. SARS-CoV-2 Receptor ACE2 Is an Interferon-Stimulated Gene in Human Airway Epithelial Cells and Is Detected in Specific Cell Subsets across Tissues. Cell. 2020 May 28;181(5):1016-1035.e19. doi: 10.1016/j.cell.2020.04.035. Epub 2020 Apr 27. PMID 32413319
- [Background] Huang J, Hume AJ, Abo KM, Werder RB, Villacorta-Martin C, Alysandratos KD, Beermann ML, Simone-Roach C, Lindstrom-Vautrin J, Olejnik J, Suder EL, Bullitt E, Hinds A, Sharma A, Bosmann M, Wang R, Hawkins F, Burks EJ, Saeed M, Wilson AA, Muhlberger E, Kotton DN. SARS-CoV-2 Infection of Pluripotent Stem Cell-Derived Human Lung Alveolar Type 2 Cells Elicits a Rapid Epithelial-Intrinsic Inflammatory Response. Cell Stem Cell. 2020 Dec 3;27(6):962-973.e7. doi: 10.1016/j.stem.2020.09.013. Epub 2020 Sep 18. PMID 32979316
- [Background] Karki R, Sharma BR, Tuladhar S, Williams EP, Zalduondo L, Samir P, Zheng M, Sundaram B, Banoth B, Malireddi RKS, Schreiner P, Neale G, Vogel P, Webby R, Jonsson CB, Kanneganti TD. Synergism of TNF-alpha and IFN-gamma Triggers Inflammatory Cell Death, Tissue Damage, and Mortality in SARS-CoV-2 Infection and Cytokine Shock Syndromes. Cell. 2021 Jan 7;184(1):149-168.e17. doi: 10.1016/j.cell.2020.11.025. Epub 2020 Nov 19. PMID 33278357
- [Background] Brodin P. Immune determinants of COVID-19 disease presentation and severity. Nat Med. 2021 Jan;27(1):28-33. doi: 10.1038/s41591-020-01202-8. Epub 2021 Jan 13. PMID 33442016
- [Background] Schuler BA, Habermann AC, Plosa EJ, Taylor CJ, Jetter C, Negretti NM, Kapp ME, Benjamin JT, Gulleman P, Nichols DS, Braunstein LZ, Hackett A, Koval M, Guttentag SH, Blackwell TS, Webber SA, Banovich NE; Vanderbilt COVID-19 Consortium Cohort; Human Cell Atlas Biological Network; Kropski JA, Sucre JM. Age-determined expression of priming protease TMPRSS2 and localization of SARS-CoV-2 in lung epithelium. J Clin Invest. 2021 Jan 4;131(1):e140766. doi: 10.1172/JCI140766. PMID 33180746
- [Background] Heiss R, Grodzki DM, Horger W, Uder M, Nagel AM, Bickelhaupt S. High-performance low field MRI enables visualization of persistent pulmonary damage after COVID-19. Magn Reson Imaging. 2021 Feb;76:49-51. doi: 10.1016/j.mri.2020.11.004. Epub 2020 Nov 18. PMID 33220447
- [Derived] Heiss R, Tan L, Schmidt S, Regensburger AP, Ewert F, Mammadova D, Buehler A, Vogel-Claussen J, Voskrebenzev A, Rauh M, Rompel O, Nagel AM, Levy S, Bickelhaupt S, May MS, Uder M, Metzler M, Trollmann R, Woelfle J, Wagner AL, Knieling F. Pulmonary Dysfunction after Pediatric COVID-19. Radiology. 2023 Mar;306(3):e221250. doi: 10.1148/radiol.221250. Epub 2022 Sep 20. PMID 36125379

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04990531/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04990531/SAP_001.pdf